CLINICAL TRIAL: NCT00111930
Title: Biological Effects of DHEA in the Elderly
Brief Title: Biological Effects of Dehydroepiandrosterone (DHEA) in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AG0019; AG018857
Record Dates: First submitted 2005-05-26; First posted 2005-05-27 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-02

CONDITIONS: Healthy
Keywords: dehydroepiandrosterone; DHEAS; bone mineral density; body composition; lean mass; fat mass; bone mass; decreased DHEAS levels
MeSH Terms: interventions — Dehydroepiandrosterone

INTERVENTIONS:
Drug: DHEA

SUMMARY:
The purpose of the study is to examine whether DHEA replacement therapy is associated with beneficial changes in body composition (i.e., increases in lean mass and bone mass, and decreases in fat mass).

DETAILED DESCRIPTION:
The central hypothesis of this study is that restoring circulating levels of the adrenal hormone dehydroepiandrosterone (DHEA) in older people with low levels to more youthful levels will be associated with beneficial changes in lean mass, fat mass and bone mass.

This will be a randomized, placebo-controlled, double-blinded study. Seventy-two men and 72 women, over 60 years old, who are healthy, will be randomized to receive either a replacement dose of DHEA or placebo for 1 year. The replacement dose of DHEA will bring circulating DHEA sulfate (DHEAS) levels into the range of normal in healthy 20-30 year-old women (approximately 8 micromoles per liter [μM] or 295 micrograms per deciliter [µg/dL]) and men (approximately 10 micromoles per liter [μM] or 368 micrograms per deciliter [µg/dL]).

Fat mass and fat-free body mass will be evaluated by dual energy x-ray absorptiometry (DXA), and intra-abdominal fat volume and thigh muscle area will be measured by computed tomography (CT). Bone mineral density (BMD) of the total body, lumbar spine, and proximal femur will be measured by DXA and biochemical markers of bone resorption and formation. Glucose tolerance and insulin response will be evaluated using an oral glucose tolerance test.

If this study confirms the results of a previous preliminary study, the current study is likely to impact future scientific study regarding the role of DHEA deficiency in the biology of aging and its role as a therapeutic agent for the prevention of sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women and men
* Age 60 or older
* Age-appropriate DHEAS levels, but 70% lower than normal DHEAS levels for a 25-year old

Exclusion Criteria:

* Contraindications to DHEA treatment (personal history of breast cancer or other estrogen-dependent neoplasms, acute liver disease, undiagnosed vaginal bleeding in women, history or evidence of prostate cancer or benign prostatic hyperplasia (BPH) in men)
* Angina
* Resting blood pressure over 180/95
* Chronic infections
* Hypothyroidism
* Depression
* Hormone therapy within the previous 6 months
* Insulin-dependent or poorly controlled diabetes
* Serum DHEAS level greater than 140 micrograms per deciliter (µg/dL)

Prohibited Medications:

* Hormone therapy other than stable regimen of thyroid replacement
* Oral glucocorticoids
* Insulin

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144
Dates: Start 2000-08; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
bone mineral density
body composition

SECONDARY OUTCOMES:
blood lipids/lipoproteins
glucose tolerance
arterial compliance
visceral adiposity
quality of life
sex steroids and growth factors
sexual health
cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Wendy M. Kohrt, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado at Denver and Health Sciences Center, Denver, Colorado, United States

REFERENCES:
- [Background] Villareal DT, Holloszy JO. Effect of DHEA on abdominal fat and insulin action in elderly women and men: a randomized controlled trial. JAMA. 2004 Nov 10;292(18):2243-8. doi: 10.1001/jama.292.18.2243. PMID 15536111
- [Background] Legrain S, Girard L. Pharmacology and therapeutic effects of dehydroepiandrosterone in older subjects. Drugs Aging. 2003;20(13):949-67. doi: 10.2165/00002512-200320130-00001. PMID 14561100
- [Background] Kahn AJ, Halloran B, Wolkowitz O, Brizendine L. Dehydroepiandrosterone supplementation and bone turnover in middle-aged to elderly men. J Clin Endocrinol Metab. 2002 Apr;87(4):1544-9. doi: 10.1210/jcem.87.4.8396. PMID 11932279
- [Background] Nippoldt TB, Nair KS. Is there a case for DHEA replacement? Baillieres Clin Endocrinol Metab. 1998 Oct;12(3):507-20. doi: 10.1016/s0950-351x(98)80286-3. PMID 10332570
- [Result] Jankowski CM, Gozansky WS, Schwartz RS, Dahl DJ, Kittelson JM, Scott SM, Van Pelt RE, Kohrt WM. Effects of dehydroepiandrosterone replacement therapy on bone mineral density in older adults: a randomized, controlled trial. J Clin Endocrinol Metab. 2006 Aug;91(8):2986-93. doi: 10.1210/jc.2005-2484. Epub 2006 May 30. PMID 16735495
- [Result] Jankowski CM, Gozansky WS, Kittelson JM, Van Pelt RE, Schwartz RS, Kohrt WM. Increases in bone mineral density in response to oral dehydroepiandrosterone replacement in older adults appear to be mediated by serum estrogens. J Clin Endocrinol Metab. 2008 Dec;93(12):4767-73. doi: 10.1210/jc.2007-2614. Epub 2008 Sep 23. PMID 18812486